CLINICAL TRIAL: NCT01305798
Title: The Effect of Time-Slot Scheduling and Active Choice on Biometric Screening Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0003; P30AG034532 (NIH)
Record Dates: First submitted 2010-11-30; First posted 2011-03-01 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Preventative Health
Keywords: Biometric Screenings; Active Choice; Behavioral Economics; Default
MeSH Terms: interventions — Appointments and Schedules

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Arm (Experimental): The control arm will be informed via e-mail of the window of dates during which they can take part in the on-site screening and will be given instructions for scheduling an appointment.
  Interventions: Other: Scheduling and Active Choice for Biometric Participation
- Active Choice and Default Option Arm (Experimental): The active choice and default option arm will be informed via e-mail of a preselected time and date for their screening, which we will have generated randomly. This group will be asked to accept the default time, schedule a different time, defer the scheduling decision, or decline to receive a screening by clicking the appropriate option in the email.
  Interventions: Other: Scheduling and Active Choice for Biometric Participation
- Active Choice Only Arm (Experimental): The active choice only arm will be given the same information as the control group, but they will also be asked to make an appointment immediately, defer the scheduling decision, or decline to receive a screening.
  Interventions: Other: Scheduling and Active Choice for Biometric Participation

INTERVENTIONS:
Other: Scheduling and Active Choice for Biometric Participation — The control group will be informed via e-mail of the window of dates during which they can take part in the on-site screening and will be given instructions for scheduling an appointment. The active choice and default option arm will be informed via e-mail of a preselected time and date for their screening, which we will have generated randomly. This group will be asked to accept the default time, schedule a different time, defer the scheduling decision, or decline to receive a screening by clicking the appropriate option in the email. The active choice only arm will be given the same information as the control group, but they will also be asked to make an appointment immediately, defer the scheduling decision, or decline to receive a screening.

SUMMARY:
The goal of this project is to see if behavioral nudges will increase an individual's likelihood of participating in a biometric screening. The behavioral nudges under consideration are assigning preselected time-slots, encouraging subjects to make an active choice, and sending reminders.

DETAILED DESCRIPTION:
The employees in our sample will schedule their time slot for a biometric screening via e-mail and a health service provider website. Much as is the case in the current system, the control group will be informed via e-mail of the window of dates during which they can take part in the on-site screening and given instructions for scheduling an appointment. The first treatment group, the active choice and default option arm, will be informed via e-mail of a preselected time and date for their screening, which we will have generated randomly. This group will be asked to accept the default time, schedule a different time, defer the scheduling decision, or decline to receive a screening by clicking the appropriate option in the email. The second treatment group, the active choice only arm, will be given the same information as the control group, but they will also be asked to make an appointment immediately, defer the scheduling decision, or decline to receive a screening. The two treatment groups will also receive email reminders one week before their appointment and again one day before their appointment.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Express Scripts
* Employee at a targeted Express Scripts location

Exclusion Criteria:

* Non-employees of Express Scripts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11000 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of employees enrolled in the intervention who complete a biometric screening through their work on-site clinic. | up to 6 months
  We will measure the employee biometric screening completion rates for each arm of the study.

CONTACTS AND LOCATIONS:
Overall Officials: David I Laibson, Ph.D, Principal Investigator — National Bureau of Economic Research
Locations (1):
- Express Scripts, St Louis, Missouri, United States